CLINICAL TRIAL: NCT05478031
Title: A Randomized, Placebo-controlled, Double-blind, Parallel-group Phase 2a Exploratory Study With Placebo run-in to Investigate PK/PD Effects, Safety, Tolerability and Pharmacokinetics of REM0046127 Oral Suspension Compared With Placebo in Subjects With Mild to Moderate Alzheimer's Disease
Brief Title: A Phase 2a Study to Investigate REM0046127 in Mild to Moderate Alzheimer's Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to the event of repeated elevated transaminase levels in one subject - elevated ALT/AST up to 6x ULN in the absence of any other potential underlying cause - we have decided to terminate the study.
Sponsor: reMYND (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REMAD-02
Record Dates: First submitted 2022-06-09; First posted 2022-07-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2024-06

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — Suspensions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- REM0046127 high dose: 1400mg (700mg bid) oral suspension (Active Comparator): REM0046127 high dose: 1400mg (700mg bid) oral suspension per day for 28 days
  Interventions: Drug: REM0046127 High Dose
- REM0046127 low dose: 350mg (175mg bid) oral suspension (Active Comparator): REM0046127 low dose: 350mg (175mg bid) oral suspension per day for 28 days
  Interventions: Drug: REM0046127 Low Dose
- Placebo (Placebo Comparator): Placebo: placebo oral suspension bid for 28 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: REM0046127 High Dose — Each subject will start with a 14-day placebo run-in period, followed by a 28-day treatment period and 7-day follow-up period.
  REM0046127 high dose: 1400mg (700mg bid) oral suspension per day for 28 days
  Other Names: 1400mg oral suspension
  Arms: REM0046127 high dose: 1400mg (700mg bid) oral suspension
Drug: REM0046127 Low Dose — Each subject will start with a 14-day placebo run-in period, followed by a 28-day treatment period and 7-day follow-up period.
  REM0046127 low dose: 350mg (175mg bid) oral suspension per day for 28 days
  Other Names: 350mg oral suspension
  Arms: REM0046127 low dose: 350mg (175mg bid) oral suspension
Drug: Placebo — Each subject will start with a 14-day placebo run-in period, followed by a 28-day treatment period and 7-day follow-up period.
  Placebo: placebo oral suspension bid for 28 days and during the 14-days run-in phase
  Other Names: 0 mg oral suspension
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure effects on CSF biomarkers, EEG and safety with REM0046127 oral suspension compared with placebo in subjects with mild to moderate Alzheimer disease.

* The study duration will be up to 2 months for each treated subject
* Each subject will start with a 14-day placebo run-in period, followed by a 28-day treatment period and 7-day follow-up period
* Visit frequency: every week
* Number of Subjects: at least 30 subjects with an upper limit of 60 subjects.
* Study Arms and Duration: All subjects will be randomized (1:1:1 allocation) to one ofthree different starting levels after the 14-day run-in period:

  * REM0046127 high dose: 1400mg (700mg bid) oral suspension per day for 28 days
  * REM0046127 low dose: 350mg (175mg bid) oral suspension per day for 28 days
  * Placebo: placebo oral suspension bid for 28 days

DETAILED DESCRIPTION:
REM0046127 is a small molecule intended for the oral treatment of subjects suffering from Alzheimer's disease (AD). The pharmacological mechanism of REM0046127 is based on modulating Orai calcium (Ca2+) channel activity to normalize neuronal Ca2+ homeostasis in ADdiseased neurons. This mechanism is central in the AD-disease cascade and is therefore expected to modulate fast-acting mechanisms like restoration of impaired synaptic function, neuronal network activity (EEG), secretion of tau into CSF and synaptic CSF biomarkers to improve cognition (symptomatic). It is also expected to influence processes with slower kinetics like brain amyloid plaques formation and neuronal cell death to slow or even stop disease progression over time (neuroprotection).

ELIGIBILITY:
Inclusion Criteria:

1. Mild to moderate AD as characterized by the following clinical, cognitive, and functional criteria.

   1. Biomarker profile reflecting AD, according to The National Institute on Aging- Alzheimer's Association (NIA-AA) Research Framework based on Screening CSF Aβ1-42 and p-tau concentrations
   2. Clear EEG deficit as assessed by the EEG reader
   3. MMSE score above 12 (preferably above 16) and a maximum of 24
2. A brain imaging study, such as magnetic resonance imaging (MRI) and/or computed tomography (CT) scan having been performed within last 6 months from day of the Screening visit or during the Screening phase of this study consistent with the clinical diagnosis of AD and excluding other potential causes of dementia. If there has been a significant change in clinical status suggestive of stroke or other possible central neurological disease with onset between the time of the last MRI or CT and the Screening evaluation, an MRI scan should be repeated during Screening procedures if considered appropriate by the Investigator
3. Age 50 to 85
4. BMI above 18 and below 35 kg/m2 (preferably below 30 kg/m2)
5. If taking concomitant medications, treated with stable doses of drugs essentially required for chronic medical conditions which do not lead to exclusion, during a period of at least 3 months prior to screening, and dose regimen is expected to remain stable during theconduct of the study
6. If taking an approved cholinesterase inhibitor or NMDA antagonist for treatment of Alzheimer's disease, treated with a stable dose for at least 6 months prior to the screening visit and the dose is not expected to change during the study as per investigators judgement, or must be off such Alzheimer medication for a period of 8 weeks prior to screening
7. Willing and able to give informed consent.
8. Have a caregiver who assists the participant every day and has intimate knowledge of the participant's cognitive, functional, and emotional states and of the participant's personal care. The caregiver must be willing to accompany the participant to all study visits and to supervise IMP administration as well as report adverse events. The caregiver must be willing and able to give informed consent for their own participation and be able to read and write.
9. Be able to read, write, speak clearly for the cognitive tests, with eyesight and hearingsufficient to enable completion of the cognitive tests

Exclusion Criteria:

1. COVID-19 positive test at the screening visit
2. Clinical, laboratory or neuro-imaging findings consistent with:

   i. Other primary degenerative dementia, (dementia with Lewy bodies, frontotemporal dementia, Huntington's disease, Creutzfeldt-Jakob Disease, Down's syndrome, etc.) ii. Other neurodegenerative condition (Parkinson's disease, amyotrophic lateral sclerosis, etc.) iii. Cerebrovascular disease (major infarct, one strategic or multiple lacunar infarcts, extensive white matter lesions > one quarter of the total white matter) iv. Other central nervous system diseases (severe head trauma, tumors, subdural hematoma or other space occupying processes, etc.) v. Seizure disorder vi. Other infectious, metabolic or systemic diseases affecting central nervous system (syphilis, present hypothyroidism, present vitamin B12 or folate deficiency, serum electrolytes out of normal range, juvenile onset diabetes mellitus, etc.)
3. Current presence of a clinically significant major psychiatric disorder according to the criteria of the DSM-IV, or symptom that could affect the subject's ability to complete the study
4. Current clinically significant systemic illness, e.g., neoplasia, that is likely to result in deterioration of the subject's condition or affect the subject's safety during the study
5. History of adrenal gland insufficiency
6. History of severe post-lumbar puncture syndrome
7. Abnormalities in the blood clotting system or abnormal coagulation status
8. Women of childbearing potential.
9. Male subjects with female partners of child-bearing potential who are unwilling or unable to adhere to contraception requirements
10. Participation in another clinical study during the last 3 months
11. Wheelchair-bound or bed-ridden
12. Any other criteria which in the opinion of the Investigator causes the subject not to qualify for the study

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Adverse Events | From first dosing to 7 days after last dose as follow-up. 14 days Run-in + 28 days treament + 7 days Follow-up
  Incidence of treatment-emergent adverse events. Number of Adverse Events either related or not related to treatment in the verum arms in comparison to the placebo arm.

CONTACTS AND LOCATIONS:
Overall Officials: Jort Vijverberg, MD, Principal Investigator — BRC Amsterdam; Koen De Witte, PhD, Study Director — CEO of reMYND
Locations (3):
- BRC Amsterdam, Amsterdam, Amsterdam, Netherlands
- Spain (2):
  - Fundacion ACE, Barcelona
  - FISEVI Hospital Universitario Virgen del Rocio, Seville

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nuytten M, Voets M, Debroux E, Princen K, Pringels L, Fivaz M, Byl E, Ramael S, De Witte K, Boada M, Morato X, Tartari JP, Lafuente A, Macias EF, Matias-Guiu JA, Vijverberg E, Teunissen CE, Anderer P, Staggs V, Hayman V, Corbett A, Ballard C, Harrison JE, Windisch M, Westman AB, Zetterberg H, Dickson S, Mallinckrodt C, Hendrix S, Cummings J, Griffioen G. Randomized phase 2a trial assessing a novel septin molecular glue in Alzheimer's disease. Alzheimers Dement. 2025 Sep;21(9):e70537. doi: 10.1002/alz.70537. PMID 40937833